CLINICAL TRIAL: NCT04049565
Title: Procalcitonin Versus C-Reactive Protein for the Guidance of Antibiotic Therapy in Critically Ill Septic Patients
Brief Title: CRP Versus PCT as Bio-markers for Sepsis and in Guiding Antibiotics in Critically Ill Patients
Acronym: PCTCRP
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Walid Ahmed Ali, Clinical Pharmacist / Walid Ahmed Ali Abdeltawab, Beni-Suef University
Other Study IDs: PCTCRP
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Sepsis; Morality
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Procalcitonin: septic patients who will receive Procalcitonin
  Interventions: Diagnostic Test: Procalcitonin biomarker and CRP biomarker
- C-Reactive Protein: septic patients who will receive C-Reactive ptotein
  Interventions: Diagnostic Test: Procalcitonin biomarker and CRP biomarker

INTERVENTIONS:
Diagnostic Test: Procalcitonin biomarker and CRP biomarker — collecting blood samples to measure serum CRP and Procalcitonin

SUMMARY:
Sepsis is a life threatening organ dysfunction caused by infection. Severe sepsis is expected to rise due to resistance to antibiotics. Inappropriate use of antibiotics in the ICU leads to adverse drug reaction and bacterial resistance. Using biomarkers for infection as PCT and CRP are useful in diagnosing infection and duration of therapy. CRP based protocol will be compared to PCT based protocol for reducing the length of stay and reduction of antibiotic use in critically ill patients.

DETAILED DESCRIPTION:
Sepsis is a syndrome of physiologic, pathologic, and biochemical abnormalities induced by infection. It is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection. It is a major public health concern, accounting for more than $20 billion (5.2%) of total US hospital costs in 2011. Not only is sepsis expensive and prevalent, but it is a major cause of mortality and critical illness worldwide. Moreover, cases of severe sepsis are expected to rise in the future for several reasons, including: Increased awareness and sensitivity for the diagnosis; increasing numbers of immunocompromised patients; wider use of invasive procedures; more resistant microorganisms; and old aging population.

Use of appropriate antibiotics in the intensive care unit (ICU) is a major challenge. Studies have shown that up to 50% of antibiotics prescribed in hospital settings are either unnecessary or inappropriate, contributing to increasing rates of resistant organisms, increases in adverse drug reactions, overall length of stay (LOS) and mortality. In addition, in critically ill patients, a long duration of treatment with antibiotics is associated with the development of antimicrobial resistance. Moreover, Sepsis and Systemic Inflammatory Response Syndrome (SIRS) SIRS can closely mimic one another and present a diagnostic challenge. So, determination of the presence or absence of bacterial infection is important to guide appropriate therapy and reduce antibiotic exposure. For microorganism detection, culture sensitivity is used though it has some drawbacks as time consuming, sometimes misleading with negative or positive reports and also they don't give information about the onset of organ dysfunction. Accordingly, it is important to differentiate culture negative sepsis patients from those with noninfectious SIRS, as these disease conditions require different therapeutic regimens. Due to these drawbacks of culture, researchers tried to depend on other more specific blood markers.

Biomarkers of infection, namely C-reactive protein and procalcitonin (PCT) have been shown to be useful in the diagnosis of infection as well as in the assessment of its response to antibiotic therapy. C-reactive protein variations overtime appears to have a good performance for the diagnosis of infection. Procalcitonin shows a better correlation with clinical severity.

Despite being used routinely in several intensive care services as an auxiliary criterion for decisions regarding antibiotic therapy, no C- reactive protein based protocol has been tested in clinical trials to guide the reduction of antibiotic use in patients with sepsis until 2012. In 2013 Oliveira et al. compared a protocol based on serum PCT levels versus a protocol based on serum C-reactive protein levels for reducing the duration of antibiotic treatment in critically ill patients presenting with severe sepsis or septic shock. The latter study showed that C-reactive protein was as useful as procalcitonin in reducing antibiotic use in a predominantly medical population of septic patients, causing no apparent harm.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 and less than 70
* Patients with sepsis or septic shock who received their first doses of antibiotics no longer than 24 h before inclusion into the study

Exclusion Criteria:

* - Elderly (defined as older than 70).
* Pregnancy and lactation
* Immunocompromised patients or who had high doses of corticosteroids
* Patients with chronic organ failure
* Infections that required long-term treatment, regardless of the etiologic agent (e.g., bacterial endocarditis).

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with sepsis or septic shock
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
compare between CRP and procalcitonin in guiding antibiotic therapy in sepsis and septic shock | one year
  measurement of the accuracy and validity of CRP and PCT as biomarkers of sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahman Dr ElNaggar, Prof, Principal Investigator — study official is dead
Locations (1):
- Cairo University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No